CLINICAL TRIAL: NCT03490448
Title: The Changes of Body Composition, Glucolipid Metabolism and Bone Metabolism in Obese Children and Adolescents After Weight Loss Camp
Brief Title: The Changes of Body Composition, Glucolipid Metabolism and Bone Metabolism in Obese Children After Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, qingya tang, chief physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: XH-DCN-Obesity
Record Dates: First submitted 2018-03-22; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Obesity, Childhood; Vitamin D Deficiency
Keywords: vitamin D; obesity; body composition; glucose metabolism; lipid metabolism
MeSH Terms: conditions — Pediatric Obesity; Vitamin D Deficiency; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Other): aerobic exercise and appropriate caloric control
  Interventions: Behavioral: aerobic exercise and appropriate caloric control

INTERVENTIONS:
Behavioral: aerobic exercise and appropriate caloric control — The dietary was designed on the basis of ensuring the daily energy physiological requirement, and basal metabolic rate (BMR) was calculated to formulate diet project according to Harris-Benedict formula. The diet was composed of 20% protein, 30% fat and 50% carbohydrates.In the exercise, heart rate was monitored to ensure the small-medial load aerobic exercise. All kinds of sports were conducted indoor, twice per day, 6 days per week, and lasted for 2 hours every time.

SUMMARY:
Vitamin D plays a significant role in calcium and phosphorus homeostasis for maintaining structural integrity and function of musculoskeletal system. Furthermore, recent studies have revealed that vitamin D can decrease the risk of many conditions other than skeletal disease, including autoimmune diseases, cancers, obesity and obesity-related diseases, such as type 2 diabetes and cardiovascular disease. Vitamin D may influence calcium absorption to affect obesity indirectly, regulate adipocyte differentiation and relieve the development of metabolic syndrome by mediating levels of inflammatory factors.

Another indicator of bone metabolism-osteocalcin may also be involved in energy metabolism and glucose metabolism, and undercarboxylated osteocalcin (ucOC) is the form which has physiological activity. ucOC may recombine with the receptors on the surface of pancreas β cells, adipocytes, hepatocytes and intestinal endocrine cell to regulate insulin secretion and insulin sensitivity.

Currently, the prevalence of vitamin D deficiency is a global problem in all age groups currently, even in countries with sun exposure all year around. The obesity group tend to have a higher incidence of vitamin D deficiency.Moreover, the obesity group tend to have a higher incidence of vitamin D deficiency and a lower level of serum osteocalcin.

This study observed the changes of body composition and glucolipid metabolism and bone metabolism during weight loss, and investigated the correlations among them.

DETAILED DESCRIPTION:
Obese children have a higher incidence of vitamin D deficiency (VDD), which resulted from unhealthy life style such as less time outdoors, more sedentary time, imbalance of dietary intake. Adipose tissue is the storage position of vitamin D, and the storage formation include 25-OHD2 and 25-OHD3. Theoretically, the reserves of vitamin D in adipose tissue of obese children might release to the circulation after weight loss. For further, it is necessary to clarify the relationship between the improvement of metabolic risk with vitamin D status after weight loss.

Osteocalcin is produced and secreted by osteoblast specifically. Recent studies have shown that it regulated glucose metabolism and energy metabolism. Obese group may have a lower level of serum osteocalcin. Both 25-OHD and osteocalcin have association with energy metabolism. This study will provide evidence to realize the relationship between bone metabolism and obesity.

In our study, all subjects were recruited from the obese children and adolescents aged 9~17 years who participated in six-week weight loss camp in July ~ August, 2014. Body mass index (BMI) was calculated as weight (kg) divided by height squared (m2). Obesity was defined as having a BMI greater than or equal to the 95th percentile for age and sex according to WHO standard. Exclusion criteria included: 1) obesity caused by endocrine or heredity diseases (eg, hypothyroidism, Prader-Willi syndrome, single-gene defects); 2) any disease influencing vitamin D metabolism (eg, such as metabolic bone diseases, rickets, nephritic syndrome and hepatic failure); 3) any supplementation use or any medication affecting vitamin D metabolism use.

All subjects underwent a closed-off weight loss program for six weeks. The intervention methods included aerobic exercise and appropriate caloric control. The dietary was designed on the basis of ensuring the daily energy physiological requirement, and basal metabolic rate (BMR) was calculated to formulate diet project according to Harris-Benedict formula. The diet was composed of 20% protein, 30% fat and 50% carbohydrates. During the camp, all subjects had never taken any kinds of nutritional supplements.

Before intervention, all subjects received exercise load test to ensure safe and effective physical exercise. In the exercise, heart rate was monitored to ensure the small-medial load aerobic exercise. The exercise programs included ball games, such as badminton, table tennis, and basketball, and also included jogging, brisk walking, swimming and cycle ergometer. All kinds of sports were conducted indoor, twice per day, 6 days per week, and lasted for 2 hours every time. The weight loss camp was staffed by professional sports coaches and medical workers. Exercise intensity was estimated by a formula: exercise intensity (target heart rate) =resting heart rate + heart rate reserve (maximum heart rate-resting heart rate) × (20%~40%).

Before and after intervention, fasting blood samples were collected and sent to Shanghai Adicon Central Lab Test Menu immediately stored in 4°C ice packs. The indicators of glucolipid metabolism and bone metabolism were tested. Total cholesterol (TC) with cholesterol oxidase, triglyceride (TG) with enzyme method (GPO-POD), high density lipoprotein (HDL) and low density lipoprotein (LDL) with homogeneous methods, fasting blood glucose (FBG) with hexokinase (HK) method, fasting insulin (FINS) with chemiluminescence method. Among the indicators of bone metabolism, osteocalcin, parathyroid hormone (PTH) and 25-OHD were assayed by electrochemiluminescence immunoassay, while bone specific alkaline phosphatase (BALP), total propeptide of type I procollagen (T-PINP) and β-isomerized form carboxy-terminal telopeptide of type I collagen (β-CTX) were determined by immunoenzymatic methods.

After blood samples were collected, anthropometric parameters were measured, including height (Seca 264, Germany), weight (Biospace 370, South Korea), triceps skinfold thickness (TST) and subscapular skinfold thickness (SST) (skinfold caliper 689900). For error reduction, every anthropometric measurement was conducted by the same trained personnels before and after weight-loss.

ELIGIBILITY:
Inclusion Criteria:

* Obesity was defined as having a body mass index (BMI) greater than or equal to the 95th percentile for age and sex according to WHO standard. BMI was calculated as weight (kg) divided by height squared (m2).

Exclusion Criteria:

* 1) obesity caused by endocrine or heredity diseases (eg, hypothyroidism, Prader-Willi syndrome, single-gene defects);
* 2) any disease influencing vitamin D metabolism (eg, such as metabolic bone diseases, rickets, nephritic syndrome and hepatic failure);
* 3) any supplementation use or any medication affecting vitamin D metabolism use.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2014-07-06 (Actual); Primary Completion 2014-08-16 (Actual); Study Completion 2014-08-16 (Actual)

PRIMARY OUTCOMES:
changes of serum 25-OHD after weight loss | after six-week weight loss camp

SECONDARY OUTCOMES:
changes of serum osteocalcin after weight loss | after six-week weight loss camp
changes of body composition after weight loss | after six-week weight loss camp
  Indicators of body composition included weight, body mass index, triceps skinfold thickness and subcutaneous skinfold thickness.
changes of glucolipid metabolism after weight loss | after six-week weight loss camp
  Indicators of glucose metabolism included fasting blood glucose (FBG) and fasting insulin (FINS). Indicators of lipid metabolism included Total cholesterol (TC), triglyceride (TG), high density lipoprotein (HDL) and low density lipoprotein (LDL).

OTHER OUTCOMES:
changes of other bone metabolism indicators after weight loss | after six-week weight loss camp
  Other bone metabolism indicators included parathyroid hormone (PTH), bone specific alkaline phosphatase (BALP), total propeptide of type I procollagen (T-PINP) and β-isomerized form carboxy-terminal telopeptide of type I collagen (β-CTX).

CONTACTS AND LOCATIONS:
Overall Officials: Qingya Tang, Mater, Principal Investigator — Department of Clinical Nutrition, Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Awad AB, Alappat L, Valerio M. Vitamin d and metabolic syndrome risk factors: evidence and mechanisms. Crit Rev Food Sci Nutr. 2012;52(2):103-12. doi: 10.1080/10408391003785458. PMID 22059957
- [Result] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Result] Holick MF. Vitamin D: importance in the prevention of cancers, type 1 diabetes, heart disease, and osteoporosis. Am J Clin Nutr. 2004 Mar;79(3):362-71. doi: 10.1093/ajcn/79.3.362. PMID 14985208
- [Result] Lee NK, Sowa H, Hinoi E, Ferron M, Ahn JD, Confavreux C, Dacquin R, Mee PJ, McKee MD, Jung DY, Zhang Z, Kim JK, Mauvais-Jarvis F, Ducy P, Karsenty G. Endocrine regulation of energy metabolism by the skeleton. Cell. 2007 Aug 10;130(3):456-69. doi: 10.1016/j.cell.2007.05.047. PMID 17693256
- [Result] Ferron M, Hinoi E, Karsenty G, Ducy P. Osteocalcin differentially regulates beta cell and adipocyte gene expression and affects the development of metabolic diseases in wild-type mice. Proc Natl Acad Sci U S A. 2008 Apr 1;105(13):5266-70. doi: 10.1073/pnas.0711119105. Epub 2008 Mar 24. PMID 18362359
- [Result] Liu JJ, Chen YY, Mo ZN, Tian GX, Tan AH, Gao Y, Yang XB, Zhang HY, Li ZX. Relationship between serum osteocalcin levels and non-alcoholic fatty liver disease in adult males, South China. Int J Mol Sci. 2013 Sep 30;14(10):19782-91. doi: 10.3390/ijms141019782. PMID 24084725
- [Result] Palacios C, Gonzalez L. Is vitamin D deficiency a major global public health problem? J Steroid Biochem Mol Biol. 2014 Oct;144 Pt A:138-45. doi: 10.1016/j.jsbmb.2013.11.003. Epub 2013 Nov 12. PMID 24239505
- [Result] Nam GE, Kim DH, Cho KH, Park YG, Han KD, Kim SM, Lee SH, Ko BJ, Kim MJ. 25-Hydroxyvitamin D insufficiency is associated with cardiometabolic risk in Korean adolescents: the 2008-2009 Korea National Health and Nutrition Examination Survey (KNHANES). Public Health Nutr. 2014 Jan;17(1):186-94. doi: 10.1017/S1368980012004855. Epub 2012 Nov 20. PMID 23168294
- [Result] Torun E, Gonullu E, Ozgen IT, Cindemir E, Oktem F. Vitamin d deficiency and insufficiency in obese children and adolescents and its relationship with insulin resistance. Int J Endocrinol. 2013;2013:631845. doi: 10.1155/2013/631845. Epub 2013 Mar 27. PMID 23606841
- [Result] Wang JW, Tang QY, Ruan HJ, Cai W. Relation between serum osteocalcin levels and body composition in obese children. J Pediatr Gastroenterol Nutr. 2014 Jun;58(6):729-32. doi: 10.1097/MPG.0000000000000243. PMID 24253362
- [Derived] Niu Y, Zhao XL, Ruan HJ, Mao XM, Tang QY. Uric acid is associated with adiposity factors, especially with fat mass reduction during weight loss in obese children and adolescents. Nutr Metab (Lond). 2020 Sep 22;17:79. doi: 10.1186/s12986-020-00500-9. eCollection 2020. PMID 32983243